CLINICAL TRIAL: NCT07342075
Title: Real-world Patient Registry Study of Cerebral Small Vessel Disease
Brief Title: Registry Study of Cerebral Small Vessel Disease
Acronym: DZM-CSVD-R
Status: Recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Prof., Dongzhimen Hospital, Beijing
Other Study IDs: 2025DZMEC-516-02
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Small Vessel Diseases; Cognitive Impairment; Diffusion Tensor Imaging
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Stool specimens from patients will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Gourp

SUMMARY:
The incidence of cerebral small vessel disease (CSVD) increases with age, affecting approximately 5% of individuals over 50 years old and nearly all individuals over 90 years old. CSVD is also the most important vascular factor contributing to cognitive decline, with 45% of dementia patients attributed to CSVD. Existing interventions are similar to secondary prevention strategies for cardiovascular and cerebrovascular diseases, and no specific therapies are currently available.

CSVD-related cognitive impairment (CSVDCI) predominantly involves attention, processing speed, and executive functions, with relatively preserved memory function, and may be accompanied by non-cognitive clinical manifestations such as gait disturbances, emotional and behavioral disorders, and bladder dysfunction. Although CSVDCI can be classified under vascular cognitive impairment (VCI), there are certain differences in its clinical manifestations.

In summary, it is necessary to develop more targeted treatments for CSVD. We attempt to establish a "symptom-tongue coating-gut microbiota-imaging" system to provide data support for the subsequent exploration of CSVD treatments based on traditional Chinese medicine (TCM) syndrome differentiation and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 50 years (including 50-year-old);
2. MRI confirmed the presence of typical imaging changes of CSVD;
3. Voluntary participation in the study and be willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Patients with acute ischemic stroke or acute intracranial hemorrhage (e.g., epidural hematoma, subdural hematoma, subarachnoid hemorrhage, intracerebral hemorrhage, etc.) or a history of cerebral infarction (non-lacunar) or intracranial hemorrhage within the past 3 months;
2. Significant non-vascular white matter lesions (e.g., multiple sclerosis, adult-onset leukoencephalopathy, metabolic encephalopathy, etc.);
3. Patients with a history of cognitive impairment due to other causes (e.g., normal pressure hydrocephalus, Alzheimer's disease, Parkinson's disease, multiple sclerosis, encephalitis, etc.);
4. Severe hepatic, renal, or cardiac insufficiency (ALT or AST >2 times the upper limit of normal, or serum creatinine >1.5 times the upper limit of normal, or New York Heart Association [NYHA] functional class III or IV);
5. Patients with psychiatric disorders that affect study medication administration and evaluation;
6. Contraindications to MRI examination (e.g., claustrophobia, presence of an implantable pacemaker, etc.);
7. Patients unable to comply with follow-up examinations or other study procedures due to residential location or other reasons;
8. Participation in other clinical trial projects.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population mainly consisted of patients from the outpatient and inpatient departments of the Department of Neurology at Dongzhimen Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montreal Cognitive Assessment (MoCA) at 6 month | 6 months
  Change from baseline in Montreal Cognitive Assessment (MoCA). Score range is 0-30. Higher score means good cognition.

SECONDARY OUTCOMES:
Change from baseline in Mini-Mental State Examination (MMSE) at 6 month | 6 months
  Change from baseline in Mini-Mental State Examination (MMSE). Score range is 0-30. Higher score means good cognition.
Changes in whole-brain fiber connectivity at 6 month | 6 months
  Measure changes in whole-brain fiber connectivity on brain MRI diffusion tensor imaging (DTI).
Change from baseline in trail making test (TMT) at 6 month | 6 months
  Change from baseline in trail making test (TMT).TMT contains TMT-A and TMT-B. Both are related to age and education. The longer the duration of both tests, the poorer the ability to concentrate, process and perform.
Change from baseline in Tinetti Performance Oriented Mobility Assessment (POMA) at 6 month | 6 months
  Change from baseline in Tinetti Performance Oriented Mobility Assessment (POMA). Score range is 0-28. Lower score means higher risk of falling.
Change from baseline in instrumental activities of daily living (IADL) at 6 month | 6 months
  Change from baseline in instrumental activities of daily living (IADL). Score range is 0-24. Higher score means better daily living.
Change from baseline in Modified Rankin Scale (mRS) at 6 month | 6 months
  Change from baseline in Modified Rankin Scale (mRS).Score range is 0-6. Higher score means greater disability.
Change from baseline in the symptom at 6 month | 6 months
  Change from baseline in the symptom. The study plans to analyze whether there are statistically significant differences in the incidence of major symptoms before and after treatment. Patient-reported outcomes (PROs) will be used to record the degree of change in patients' symptoms from baseline (expressed as a percentage, with >100% indicating symptom worsening and <100% indicating symptom relief). Meanwhile, baseline and 6-month tongue coating photos will be preserved.
Change from baseline in gut microbiota at 6 month | 6 months
  Change from baseline in gut microbiota. Metagenomic sequencing technology will be applied to the analysis.

OTHER OUTCOMES:
Numbers in new vascular events from baseline to 6 month | 6 months
  New vascular events include ischemic stroke, TIA, cerebral hemorrhage, MI, pulmonary embolism, thrombosis, peripheral arterial occlusion
Numbers in all-cause hospitalization from baseline to 6 month | 6 months
  Numbers in all-cause hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, 100700, Beijing, Beijing Municipality, China